CLINICAL TRIAL: NCT06720298
Title: CD147 Targeting Peptide Probe for PET Imaging in Solid Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2024YJZ142
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor
Keywords: Solid Cancer; CD147; PET imaging
MeSH Terms: interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 68Ga-DOTA-AP9: All enrolled participants will be allocated to this arm (single-arm study). Study participants will undergo 68Ga-DOTA-AP9 PET/CT scan.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — All study participants will undergo one 18F-FDG PET/ CT scan.

SUMMARY:
The objective of the study is to construct a noninvasive approach using 68Ga-DOTA-AP9 PET/CT to detect the CD147 expression of tumor lesions in patients with solid tumors and to identify patients benefiting from CD147 targeting treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Malignant melanoma, liver cancer, colon cancer, pancreatic cancer, breast cancer, gastric cancer, lung cancer, etc., confirmed by histopathology or cytology;
2. age ≥18 and ≤75 years old, male or female;
3. ECOG score 0 or 1;
4. expected survival time ≥6 months;
5. There was at least one measurable target lesion according to RECIST1.1 criteria, and biopsy could be performed within one month before and after PET scan, and the patient could provide 2-3 lesion tissue slides;
6. Women of childbearing age (15-49 years) must have had a negative pregnancy test within 7 days before starting testing; Women and men of childbearing potential must agree to use effective contraception to avoid pregnancy during the study and for 3 months after the examination;
7. patients recommended by clinicians to undergo PET/CT examination for tumor staging;
8. The subjects could fully understand and voluntarily participate in this experiment, and signed an informed consent.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or women planning to become pregnant during the study or within three months after administration, as well as individuals donating sperm or oocytes.
2. Individuals known or suspected to be allergic to the investigational drug or any of its components.
3. Individuals with significantly abnormal liver or kidney function: serum total bilirubin (TBIL) > 1.5 × 20 µmol/L, or aspartate aminotransferase (AST) > 2.5 × 45 µmol/L, or alanine aminotransferase (ALT) > 2.5 × 40 µmol/L, or serum creatinine > 1.5 × 130 µmol/L.
4. Unable to cooperate in completing the PET scan, or suffering from claustrophobia or other conditions that prevent cooperation during the PET scan.
5. Other situations deemed inappropriate for participation in the trial by the investigator. Female patients who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Malignant tumor patients or suspected patients
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value（SUV） | 2 years
  SUV is a semi-quantitative analysis index to describe the radioactive uptake of lesions, which has certain reference value for differentiating benign and malignant lesions. The uptake of the tracer （68Ga-DOTA-AP9） in solid tumor lesions by measuring SUV on PET/CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No